CLINICAL TRIAL: NCT01676142
Title: Establishing a Diagnostic Test for Non-tuberculous Mycobacteria Lung Infection Using Non-tuberculous Mycobacteria Antigen Stimulation Test: From Immune Base, Standardized Setup to Validation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201012082RC
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2011-06

CONDITIONS: To Set up NTM Stimulation Test Foar Diagnosing NTM Pulmonary Infectionon.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with NTM pulmonary infection
- Patients with other pathogen related lung infection
- Patient with NTM pulmonary colonization

SUMMARY:
1. To compare TLR-2 expression of peripheral blood mononuclear cells and serum downstream cytokines in those with MAC or MAB pulmonary infection and those with MAC or MAB pulmonary colonization and controls.
2. To investigate the response of TLR-2 expression and cytokines activation to NTM stimulation test in patients with MAC or MAB pulmonary infection and colonization and controls.
3. To validate the NTM stimulation test for NTM pulmonary infection.

DETAILED DESCRIPTION:
The increase of nontuberculous mycobacteria lung infection Nontuberculous mycobacteria lung infection (NTM-LD) becomes an important clinical concern [1] because the rate of NTM infection has increased over the past ten years [2-3]. According to a study in Taiwan, NTM-LD increased from 1.26 to 7.94 per 100,000 inpatients/year during 2000 to 2008 [2]. The reasons for this increase are not readily clear, but could be related to the growth in numbers of the acquired immunocompromised population and advances of technique for mycobacterial culture [4-7]. Among the NTM infection in Taiwan, Mycobacterium avium complex (MAC) and M. abscessus (MAB) were most frequently isolated [2].

The difficulty in early diagnosing and confirming true NTM-LD However, NTM exists in the environment ubiquitously, so the relevance (true disease patient number over the number of patients with disease or just colonization) is far less than 100% and varied in different NTM species. For example, previous studies have shown that the presence of M. kansasii and MAC had a clinical relevance around 47~70% and 35~42%, respectively [8-9]. As for MAB which is emerging pathogen worldwide, has a relevance of 33% [9]. According to contemporary NTM guidelines established by American thoracic society, NTM pulmonary infection is diagnosed by multiple criteria including microbiology of respiratory specimen and clinical findings as well as radiographic findings [1]. In microbiology criteria, two or more sets of positive sputum mycobacterial culture for the same NTM species within one year is needed.

Because NTM colonization is not uncommon in respiratory tract, diagnosis of true pulmonary NTM infection is a great challenge in clinical practice. Actually, microbiology tests for mycobacteria are neither timely nor efficient. Mycobacterial culture is time-consuming, which needed weeks to wait the results even though it's current gold standard for micro-organism identification [10]. The nucleic acid amplification method such as polymerase chain reaction could not discriminate true NTM infection and solely colonization because the micro-organism is present in both situations [11].

To early diagnose and then start treatment of NTM infection is important because NTM pulmonary infection might be rapid lethal infection in intensive care unit or in patients who had not received early proper treatment [6]. In addition, MAC or MAB which are most common in Taiwan are resistant to most of anti-tuberculosis regimen. Hence, more rapid and accurate diagnostic test should be developed [1-2, 6] The help of innate immunity in diagnosing NTM-LD The body inflammatory marker, represent our immune response, would be an indicator for differentiating true mycobacterial pulmonary infection from colonization while the first set of mycobacterial culture grew NTM [12-15]. Both interferon-gamma and tumor necrosis factor-alpha play critical roles in protective immunity to mycobacterial infections [16-17]. These responses are linked to engagement of Toll-like receptor 2 (TLR2) that is critical for mycobacterial infection [18]. However, the TLR-2 expression has not been evaluated between patients with NTM infection and colonization. According to the success of application of interferon-gamma release assay for tuberculosis detection [19], we understand the specific immune response is helpful to diagnose mycobacterial infection. We therefore focus on the expression of TLR-2 and associated downstream cytokines in our patients with MAC or MAB lung disease, which accounts the most of NTM infection [2].

The design in our study for diagnosis In order to investigate the help of host immune in diagnosing NTM pulmonary infection, we initially compare the baseline expression of TLR-2 and downstream cytokines in the MAC or MAB infected patients and colonized subjects. Then, we perform an in-vitro stimulation test using mycobacteria (MAC or MAB) for co-culturing with peripheral blood mononuclear cells of patients. The TLR-2 expression and cytokines activation will be examined after the stimulation test. We then analyze the expression difference between NTM-LD and colonization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A patient has at least 3 sets of respiratory specimen for mycobacterial culture.

Exclusion Criteria:

* Age younger than 18 years.
* Patients who have pregnancy.
* Patients who have acquired immunodeficiency syndrome
* Patients who have bleeding tendency which can not tolerate venous puncture such as hemophilia, thrombocytopenia.
* In NTM infection group, patients having received anti-NTM treatment for one week will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with NTM pulmonary infection: diagnosed by NTM guidelines by American Thoracic Society(ATS)
  2. Patients with NTM pulmonary colonization: Patients are not fulfilling the ATS diagnostic criteria but having at least one set of positive sputum for NTM (colonization).
  3. Patients have pulmonary infiltrates, not related by NTM: three sets of respiratory specimens that are negative for NTM.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Patients with non-tuberculous pulmonary infection | 3 year

SECONDARY OUTCOMES:
mortality | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan